CLINICAL TRIAL: NCT03388281
Title: Morbidity, Mortality and Gender Differences in Patients With Pacemakers; a Large-scale Single-center Cohort Study
Brief Title: Morbidity, Mortality and Gender Differences in Patients With Pacemakers
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Mariann Gyongyosi, Cardiologist, Assoc. Prof. Univ.-Doz. Dr., Medical University of Vienna
Other Study IDs: EK1525/2015
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Pacemaker, Artificial; Cohort Studies; Arrhythmias Requiring Therapy; Cardiac Pacing, Artificial
Keywords: Pacemaker; Gender differences; Survival; Retrospective

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with implanted pacemaker: Patients with implanted cardiac pacemaker registered in pacemaker database of the Department of Cardiology at the Medical University Vienna were included.
  Interventions: Other: No intervention, retrospective analysis only.

INTERVENTIONS:
Other: No intervention, retrospective analysis only. — No intervention, retrospective analysis only.

SUMMARY:
Previous publications suggest gender difference in outcome parameters after pacemaker implantation. Aim of this study is to investigate gender differences in patients with pacemaker. Implanted devices, indication for implantation and pacemaker follow up data of patients will be included. Survival data including cause of death will be documented. Prevalent comorbidities and relevant laboratory data will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients registered in the pacemaker database of the Department of Cardiology at the Medical University Vienna. Patients get registered when clinical follow up of an implanted Pacemaker is done.

Exclusion Criteria:

* For survival analysis: No valid match of first name AND surname AND date of birth with patients' insurance data.
* For analysis of comorbidities: Not a single documented diagnose was found in our electronic clinic-wide patients' information system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women and men with implanted cardiac Pacemaker and at least one follow up in our Pacemaker Office of the Department of Cardiology at the Medical University Vienna. Patients were enrolled regardless of time and place of pacemaker implantations.
Sampling Method: Non-Probability Sample
Enrollment: 11444 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Survival after pacemaker implantation | 10 years
  Null hypothesis: There is no survival difference between women and men after pacemaker Implantation.

SECONDARY OUTCOMES:
Implantation rates of single- or dual-chamber Pacemaker in women/men. | Data obtained: April 30th, 2015
  Null hypothesis: Women and men have equal implantation rates of single- and dual-chamber pacemakers.
Survival of women/men after single- or dual-chamber pacemaker implantation. | 10 years
  Null hypothesis: Survival after single- or dual-chamber pacemaker implantation is equal.

OTHER OUTCOMES:
First implantation age in single- or dual-chamber pacemaker | Data obtained: April 30th, 2015
  Null hypothesis: There is no difference in first implantation age between sexes and single- or dual-chamber pacemakers.
Time to device- or lead-replacement | 10 years
  Null hypothesis: There is no difference between women and men in time to device- or lead-replacement.
Prevalence of Comorbidities | Survival analysis: 10 years; data obtained: March 2nd, 2016
  Null hypothesis: There is no difference in survival and first pacemaker implantation when selected comorbidity was found.
Survival and device/lead-replacement in patients with diabetes. | 10 years
  Null hypothesis: There is no difference in survival or device/lead-replacement rates in women/men with diabetes.
Pacemaker parameters | Data obtained: April 30th, 2015
  Null hypothesis: There is no difference between women and men in pacing threshold and lead impedance.
Laboratory results | Data obtained: March 2nd, 2016
  Null hypothesis: There is no difference between women and men in troponin T, N-terminal pro-brain natriuretic Peptide, HbA1c and low-density lipoprotein.

CONTACTS AND LOCATIONS:
Overall Officials: Mariann Gyöngyösi, MD, PhD, Principal Investigator — Medical University of Vienna

IPD SHARING:
Plan to Share IPD: Yes
Sharing of IPD is planned.

REFERENCES:
- [Derived] Riesenhuber M, Spannbauer A, Rauscha F, Schmidinger H, Boszotta A, Pezawas T, Schukro C, Gwechenberger M, Stix G, Anvari A, Wrba T, Khazen C, Andreas M, Laufer G, Hengstenberg C, Gyongyosi M. Sex Differences and Long-Term Outcome in Patients With Pacemakers. Front Cardiovasc Med. 2020 Sep 22;7:569060. doi: 10.3389/fcvm.2020.569060. eCollection 2020. PMID 33195457